CLINICAL TRIAL: NCT04537312
Title: Prospective Pilot Study of Robot-Assisted Nipple Sparing Mastectomy (RNSM)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Sara Myers, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OSU-19199; NCI-2020-05349 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-08-18; First posted 2020-09-03 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Ductal Breast Carcinoma In Situ; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prophylactic Mastectomy
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Supportive care (RNSM, surveys) (Experimental): RNMS Surveys
  Interventions: Procedure: Robot-assisted Nipple Sparing Mastectomy; Other: Survey Administration; Device: RNSM

INTERVENTIONS:
Procedure: Robot-assisted Nipple Sparing Mastectomy — Under RNSM
Other: Survey Administration — ancillary correlative
Device: RNSM — Robot-assisted Nipple Sparing Mastectomy

SUMMARY:
This is a pilot study to determine safety, efficacy, and potential risks of robot assisted nipple sparing mastectomy (RNSM), by utilizing the daVinci surgical system.

DETAILED DESCRIPTION:
With the advances of breast reconstruction after mastectomy for the treatment of breast diseases including breast cancer, surgical techniques have evolved to preserve the skin flaps and nipple areolar complex (NAC) to give better aesthetic outcome without compromising outcome. Mastectomy that preserves the NAC is called nipple sparing mastectomy (NSM). NSM can provide major psychosocial benefits for patients but is technically demanding and challenging to perform. Total mammary glandular excision in NSM can be technically challenging due to small size of the incision and poor visualization of dissection plane. Recent studies demonstrate feasibility and safety of performing minimally invasive robot-assisted NSM (RNSM). The technique of RNSM is still novel.

This is a single-arm pilot study for feasibility and safety of RNSM.

ELIGIBILITY:
Inclusion Criteria:

* Surgical candidates, per standard of care for:

  * Nipple sparing resection and reconstruction OR
  * Prophylactic mastectomy for risk reduction mastectomy OR
  * Treatment of ductal carcinoma in-situ or clinically node negative cT1-T3 breast cancer
* Surgical candidates for open NSM, per standard of care, with regards to patient anatomic factors and tumor location
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Pregnant or nursing women
* Patients with:

  * Inflammatory breast cancer
  * Skin involvement with tumor
  * Pre-operative diagnosis (radiological or pathologic) of nipple-areola complex involvement with tumor
  * Grade 3 ptosis of nipple
* Smokers with heavy current use of nicotine (defined as > 20 cigarettes/day)
* Patients that are high risk for anesthesia, as documented in medical record
* Patients that do not have the ability to give informed consent
* Prisoner status at surgical clinic visit
* Bra cup size greater than C cup
* Previous thoracic radiation history (for any reason)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of removal of breast gland en bloc through RNSM | Up to 1 year
  Measure number of patients who had breast removed en bloc through RNSM incision.
Complication rate of patients with bleeding requiring re-operation | Up to 1 year
  Number of patients with bleeding requiring re-operation after RNSM.
Complication rate of patients with infection requiring antibiotics or re-operation | Up to 1 year
  Number of patients with infection after surgery requiring antibiotics or re-operation.
Complication rate of patients with Mastectomy flap (SKIN flap score) | Up to 1 year
  Number of patients with mastectomy flap or nipple-areolar complex necrosis as measured using the SKIN flap score after surgery. Score of A1 indicates normal skin, D4 indicates total full thickness necrosis.
Perioperative Outcomes investigating the total duration of surgical time | Up to 1 year
  Investigate the total duration of the operation (surgical time data),
Perioperative Outcomes investigating length of surgery time | Up to 1 year
  Investigate the total duration of the operation (surgical time data) of each patient
Perioperative Outcomes investigating the length of hospitalization | Up to 1 year
  Investigate the length of hospitalization for each patient

SECONDARY OUTCOMES:
Surgeon musculoskeletal fatigue with RNSM using (SURG-TLX) survey | Up to 1 year
  Surgery Task Load Index (SURG-TLX) survey from each surgeon performing surgery.
Surgeon musculoskeletal fatigue with RNSM using NMSQ questionnaire | Up to 1 year
  Musculo-Skeletal Questionnaire (NMSQ) from each surgeon performing surgery.
Patient Reported Outcomes | Up to 1 year
  Monofilament testing to test for sensation recovery after surgery from each participant. Semmes Weinstein monofilament exam; sensation to series of monofilament with different thickness, compare sensation to preoperative exam.
Patient Reported Outcomes | Up to 1 year
  Patient satisfaction with the breast after surgery measured by BREAST-Q survey. Lowest score = 0, highest = 100 with higher scores indicating better outcomes / quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: William Carson, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park KU, Lee S, Sarna A, Chetta M, Schulz S, Agnese D, Grignol V, Carson W, Skoracki RJ. Prospective pilot study protocol evaluating the safety and feasibility of robot-assisted nipple-sparing mastectomy (RNSM). BMJ Open. 2021 Nov 15;11(11):e050173. doi: 10.1136/bmjopen-2021-050173. PMID 34782341
- See also: The Jamesline — http://cancer.osu.edu